CLINICAL TRIAL: NCT00003099
Title: Phase II Clinical Trial of N-(4-hydroxyphenyl) Retinamide (4-HPR) and Tamoxifen in Breast Neoplasia, Administration During the Period Between the Diagnostic Core Biopsy and Definitive Surgery
Brief Title: Chemoprevention Therapy Plus Surgery in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ID94-029; P30CA016672 (NIH); MDA-ID-94029 (Other: UT MD Anderson Cancer Center); NCI-P97-0113; CDR0000065829 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; Tamoxifen; Fenretinide; Chemoprevention Therapy; N-(4-hydroxyphenyl) Retinamide; 4-HPR; Breast Neoplasia; Diagnostic Core Biopsy; Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Fenretinide; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Tamoxifen + Fenretinide (Active Comparator): Tamoxifen + Fenretinide daily for 14-28 days
  Interventions: Drug: Fenretinide; Drug: Tamoxifen Citrate
- Arm 2 Placebo (Placebo Comparator): Placebo daily for 14-28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenretinide — Daily for 14-28 days.
  Other Names: 4-HPR; N-(4-hydroxyphenyl) Retinamide
  Arms: Arm 1 Tamoxifen + Fenretinide
Drug: Tamoxifen Citrate — Daily for 14-28 days.
  Other Names: Nolvadex
  Arms: Arm 1 Tamoxifen + Fenretinide
Other: Placebo — Daily for 14-28 days
  Arms: Arm 2 Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of fenretinide and tamoxifen before surgery may be an effective way to prevent the recurrence of or further development of breast cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of fenretinide and tamoxifen given before surgery in treating women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of identifying surrogate endpoint biomarkers in women with breast ductal carcinoma in situ and associated neoplastic and preneoplastic lesions. II. Determine whether treatment with fenretinide and tamoxifen administered daily will cause significant modulation of proposed surrogate endpoint biomarkers in this patient population.

OUTLINE: This is a randomized, placebo controlled study. Patients are stratified according to histological diagnosis (hyperplasia vs carcinoma). All patients undergo a core biopsy and fine needle aspiration of the index lesion and are then assigned randomly to a treatment arm. Arm I receives tamoxifen and fenretinide daily. Arm II receives a placebo daily. Both arms continue for 14-28 days, until definitive surgery or a second biopsy is performed.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study, 50 patients per arm.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Mammogram highly suspicious for ductal carcinoma in situ or early invasive carcinoma Branching or linear microcalcifications clustered or distributed segmentally in the breast without an associated palpable or mammographic mass Palpable thickening or nipple discharge allowed At least 5 mm area of calcification or contain enough calcium for core biopsies Small palpable carcinoma (T1 or T2) with no palpable axillary lymph nodes (N0) No definitive local therapy Atypical hyperplasia (ductal or lobular) and/or carcinoma on initial diagnostic biopsy Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Over 18 Sex: Female Menopausal status: Not specified Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No uncontrolled congestive heart failure Other: Fasting serum triglycerides less than 400 mg/dL Fertile patients must use effective contraception during and for one year after completing fenretinide therapy No concurrent serious illness or infection, e.g., septicemia No prior thromboembolic disease No prior degenerative retinal disease

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 5 years since prior chemotherapy Endocrine therapy: At least 12 months since prior tamoxifen therapy No concurrent estrogen therapy At least 3 months since prior anabolic steroids Radiotherapy: No prior radiotherapy to the chest or breast Surgery: See Disease Characteristics Other: No vitamin A supplementation greater than 25,000 IU At least 12 months since prior retinoid therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 1996-05; Primary Completion 2000-06 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Fenretinide + Tamoxifen effectiveness given before surgery in treating breast cancer | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sonja E. Singletary, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org